CLINICAL TRIAL: NCT00871598
Title: A Multiple Ascending Dose Study to Assess the Safety and Pharmacokinetics of Repeated Intravenous Doses of BTT-1023 in Patients With Plaque Psoriasis - a Double-blind Randomized Placebo-controlled Sequential Group Trial
Brief Title: BTT1023 in Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biotie Therapies Corp. (Industry)
Responsible Party: CMO, Biotie Therapies, Biotie Therapies Corp.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTT12-CD016
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; BTT1023; safety; pharmacokinetics
MeSH Terms: interventions — timolumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Single 0.3 (Experimental)
  Interventions: Drug: BTT1023
- Repeat 1.0 (Experimental)
  Interventions: Drug: BTT1023
- Repeat 2.0 (Experimental)
  Interventions: Drug: BTT1023
- Repeat 4.0 (Experimental)
  Interventions: Drug: BTT1023
- Repeat 8.0 (Experimental)
  Interventions: Drug: BTT1023

INTERVENTIONS:
Drug: BTT1023 — intravenous, three infusions over three weeks
  Arms: Repeat 1.0; Repeat 2.0; Repeat 4.0; Repeat 8.0
Drug: Placebo — intravenous, three infusions over three weeks
  Arms: Placebo
Drug: BTT1023 — Test challenge
  Arms: Single 0.3

SUMMARY:
Patients with plaque psoriasis will be enrolled. They will be dosed with repeated intravenous doses of BTT-1023 or placebo. During the trial, the safety of the treatments and the pharmacokinetics of BTT-1023 will be assessed. The patient allocation to treatment groups will occur at random, and the actual treatment will not be revealed to the investigator or to the patient during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis affecting at least 8% of the body surface area and scoring 8 or higher in the psoriasis area and severity index

Exclusion Criteria:

* Seropositive for infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus; Tuberculosis; Acute systemic infection;
* Treatment with a monoclonal antibody therapy within 12 weeks prior to study entry;
* An absolute indication for a known effective treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 weeks
Plasma concentrations of BTT1023 | 12 weeks

SECONDARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Biotie investigational site, Dresden, Dresden
  - Biotie investigational site, Leipzig, Leipzig
  - Biotie investigational site, Berlin, State of Berlin
  - Biotie Investigational Site, Görlitz